CLINICAL TRIAL: NCT01121536
Title: A 6-Month, Open-Label, Flexible-Dosage (150 to 200 mg/Day) Extension Study of the Safety and Efficacy of Armodafinil Treatment as Adjunctive Therapy in Adults With Major Depression Associated With Bipolar I Disorder
Brief Title: Extension Study of the Safety and Efficacy of Armodafinil Treatment as Adjunctive Therapy in Adults With Major Depression Associated With Bipolar I Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision related to efficacy rather than tolerability limitations, not stopped for any safety reasons.
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C10953/3074; 2009-016648-38 (EudraCT Number)
Record Dates: First submitted 2010-05-05; First posted 2010-05-12 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Depression
Keywords: Bipolar I Disorder
MeSH Terms: conditions — Depression | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Armodafinil 150-200 mg/day (Experimental): Participants began taking armodafinil at a dosage of 50 mg/day; the dosage was increased by 50 mg/day on days 2 and 4, up to a dosage of 150 mg/day. At the discretion of the investigator, the dosage of armodafinil may be increased to 200 mg/day on day 6 or thereafter, and reduced to 150mg/day if the higher dose is not well tolerated. Treatment was administered for six months.
  Interventions: Drug: Armodafinil

INTERVENTIONS:
Drug: Armodafinil — Armodafinil tablets, taken orally, once daily in the morning
  Other Names: CEP-10953; Nuvigil

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of long term (6 months) armodafinil treatment as adjunctive therapy to mood-stabilizing medications in adults with bipolar I disorder.

ELIGIBILITY:
Key Inclusion Criteria:

* The patient has completed 8 weeks of treatment in a Cephalon-sponsored Phase 3, double-blind study of armodafinil treatment in patients with major depression associated with bipolar I disorder.
* The patient met criteria for enrollment in the previous double-blind study and, in the opinion of the investigator, is in need of continued treatment for depression.
* During the previous double-blind study, the patient must have been taking 1 (or 2) of the following protocol-allowed mood stabilizers: lithium; valproic acid; olanzapine; quetiapine; aripiprazole; lamotrigine; risperidone; ziprasidone, (only if taken in combination with lithium, valproic acid, or lamotrigine). The following criteria must also be met:

  1. The mood stabilizers must be taken in an oral formulation, with the exception of risperidone, which can be either in an oral or long-acting injection formulation.
  2. The patient may be taking 2 protocol-allowed mood stabilizers only if 1 of the drugs is lithium, valproic acid, or lamotrigine.
  3. The patient must be judged by the investigator to be compliant with treatment with the mood stabilizer(s).
  4. The patient must be willing to continue treatment with the same protocol-allowed mood stabilizer(s) at dosages considered appropriate by the investigator.
* The patient has a Young Mania Rating Scale (YMRS) total score of 14 or less at the enrollment visit. Patients who have a YMRS score of 12 through 14 must be discussed with the medical monitor to determine their suitability for enrollment.

Key Exclusion Criteria:

* The patient has any Axis I or Axis II disorder apart from bipolar I disorder that became the primary focus of treatment during the double-blind study.
* The patient has psychotic symptoms or had psychosis during the double-blind study.
* The patient has current active suicidal ideation, is at imminent risk of self harm, or has a history of significant suicidal ideation or suicide attempt at any time in the past that causes concern at present.
* The patient met criteria for alcohol or substance abuse or dependence (with the exception of nicotine dependence) during the double-blind study.
* The patient has any history of homicidal ideation or significant aggression or currently has homicidal or significant aggressive ideation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 867 (Actual)
Dates: Start 2010-04-30 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2013-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (158):
- United States (66):
  - Teva Investigational Site 113, Birmingham, Alabama
  - Teva Investigational Site 225, Birmingham, Alabama
  - Teva Investigational Site 229, Anaheim, California
  - Teva Investigational Site 217, Cerritos, California
  - Teva Investigational Site 223, Cerritos, California
  - Teva Investigational Site 115, Garden Grove, California
  - Teva Investigational Site 121, Imperial, California
  - Teva Investigational Site 303, Oceanside, California
  - Teva Investigational Site 400, Oceanside, California
  - Teva Investigational Site 200, Pico Rivera, California
  - Teva Investigational Site 128, San Diego, California
  - Teva Investigational Site 201, San Diego, California
  - Teva Investigational Site 192, Santa Ana, California
  - Teva Investigational Site 292, Santa Ana, California
  - Teva Investigational Site 295, Sherman Oaks, California
  - Teva Investigational Site 122, Temecula, California
  - Teva Investigational Site 131, Gainesville, Florida
  - Teva Investigational Site 132, Jacksonville, Florida
  - Teva Investigational Site 606, Jacksonville Beach, Florida
  - Teva Investigational Site 127, Lauderhill, Florida
  - Teva Investigational Site 119, North Miami, Florida
  - Teva Investigational Site 118, Tampa, Florida
  - Teva Investigational Site 608, Tampa, Florida
  - Teva Investigational Site 205, Atlanta, Georgia
  - Teva Investigational Site 116, Atlanta, Georgia
  - Teva Investigational Site 204, Smyrna, Georgia
  - Teva Investigational Site 107, Naperville, Illinois
  - Teva Investigational Site 301, Naperville, Illinois
  - Teva Investigational Site 219, Oakbrook Terrace, Illinois
  - Teva Investigational Site 195, Park Ridge, Illinois
  - Teva Investigational Site 600, Lafayette, Indiana
  - Teva Investigational Site 300, Pikesville, Maryland
  - Teva Investigational Site 603, Watertown, Massachusetts
  - Teva Investigational Site 290, Flowood, Mississippi
  - Teva Investigational Site 133, St Louis, Missouri
  - Teva Investigational Site 103, Mount Laurel, New Jersey
  - Teva Investigational Site 212, Mount Laurel, New Jersey
  - Teva Investigational Site 193, Albuquerque, New Mexico
  - Teva Investigational Site 207, Brooklyn, New York
  - Teva Investigational Site 104, Brooklyn, New York
  - Teva Investigational Site 202, New York, New York
  - Teva Investigational Site 129, Rochester, New York
  - Teva Investigational Site 411, Staten Island, New York
  - Teva Investigational Site 110, Staten Island, New York
  - Teva Investigational Site 105, Raleigh, North Carolina
  - Teva Investigational Site 190, Beachwood, Ohio
  - Teva Investigational Site 213, Canton, Ohio
  - Teva Investigational Site 610, Cincinnati, Ohio
  - Teva Investigational Site 102, Dayton, Ohio
  - Teva Investigational Site 401, Oklahoma City, Oklahoma
  - Teva Investigational Site 609, Oklahoma City, Oklahoma
  - Teva Investigational Site 616, Oklahoma City, Oklahoma
  - Teva Investigational Site 406, Allentown, Pennsylvania
  - Teva Investigational Site 117, Media, Pennsylvania
  - Teva Investigational Site 106, Memphis, Tennessee
  - Teva Investigational Site 111, Austin, Texas
  - Teva Investigational Site 403, DeSoto, Texas
  - Teva Investigational Site 612, Friendswood, Texas
  - Teva Investigational Site 228, Houston, Texas
  - Teva Investigational Site 224, Irving, Texas
  - Teva Investigational Site 409, Orem, Utah
  - Teva Investigational Site 408, Salt Lake City, Utah
  - Teva Investigational Site 404, Richmond, Virginia
  - Teva Investigational Site 100, Bellevue, Washington
  - Teva Investigational Site 613, Kirkland, Washington
  - Teva Investigational Site 605, Spokane, Washington
- Argentina (13):
  - Teva Investigational Site 237, Buenos Aires
  - Teva Investigational Site 450, Buenos Aires
  - Teva Investigational Site 881, Buenos Aires
  - Teva Investigational Site 884, Buenos Aires
  - Teva Investigational Site 136, Buenos Aires
  - Teva Investigational Site 134, Buenos Aires
  - Teva Investigational Site 235, Buenos Aires
  - Teva Investigational Site 462, Buenos Aires
  - Teva Investigational Site 135, Córdoba
  - Teva Investigational Site 236, Córdoba
  - Teva Investigational Site 371, La Plata
  - Teva Investigational Site 138, La Plata, Buenos Aires
  - Teva Investigational Site 238, Rosario
- Australia (2):
  - Teva Investigational Site 141, Brisbane
  - Teva Investigational Site 240, Malvern
- Teva Investigational Site 624, Rio de Janeiro, Brazil
- Bulgaria (14):
  - Teva Investigational Site 248, Burgas
  - Teva Investigational Site 146, Kardzhali
  - Teva Investigational Site 148, Kazanlak
  - Teva Investigational Site 853, Pazardzhik
  - Teva Investigational Site 852, Pleven
  - Teva Investigational Site 249, Plovdiv
  - Teva Investigational Site 145, Plovdiv
  - Teva Investigational Site 370, Rousse
  - Teva Investigational Site 147, Sofia
  - Teva Investigational Site 854, Sofia
  - Teva Investigational Site 855, Sofia
  - Teva Investigational Site 247, Sofia
  - Teva Investigational Site 851, Varna
  - Teva Investigational Site 245, Varna
- Canada (4):
  - Teva Investigational Site 198, Kelowna
  - Teva Investigational Site 296, Mississauga
  - Teva Investigational Site 196, Mississauga
  - Teva Investigational Site 299, Penticton
- Croatia (3):
  - Teva Investigational Site 635, Rijeka
  - Teva Investigational Site 633, Zagreb
  - Teva Investigational Site 634, Zagreb
- France (2):
  - Teva Investigational Site 286, Dole
  - Teva Investigational Site 153, Nîmes
- Germany (2):
  - Teva Investigational Site 655, Achim
  - Teva Investigational Site 651, Dresden
- Hungary (4):
  - Teva Investigational Site 661, Budapest
  - Teva Investigational Site 664, Budapest
  - Teva Investigational Site 662, Budapest
  - Teva Investigational Site 666, Nagykálló
- Italy (4):
  - Teva Investigational Site 688, Catania
  - Teva Investigational Site 689, Florence
  - Teva Investigational Site 687, Pisa
  - Teva Investigational Site 692, Rome
- Poland (9):
  - Teva Investigational Site 259, Bialystok
  - Teva Investigational Site 258, Gdansk
  - Teva Investigational Site 257, Gdansk
  - Teva Investigational Site 156, Kielce
  - Teva Investigational Site 155, Krakow
  - Teva Investigational Site 256, Leszno
  - Teva Investigational Site 255, Skorzewo
  - Teva Investigational Site 861, Szczecin
  - Teva Investigational Site 157, Tuszyn
- Serbia (8):
  - Teva Investigational Site 832, Belgrade
  - Teva Investigational Site 175, Belgrade
  - Teva Investigational Site 177, Belgrade
  - Teva Investigational Site 831, Belgrade
  - Teva Investigational Site 833, Belgrade
  - Teva Investigational Site 176, Kragujevac
  - Teva Investigational Site 837, Niš
  - Teva Investigational Site 834, Novi Kneževac
- Slovakia (4):
  - Teva Investigational Site 699, Bratislava
  - Teva Investigational Site 697, Rimavská Sobota
  - Teva Investigational Site 696, Rožňava
  - Teva Investigational Site 698, Trenčín
- South Africa (6):
  - Teva Investigational Site 712, Cape Town
  - Teva Investigational Site 709, Cape Town
  - Teva Investigational Site 708, Centurion
  - Teva Investigational Site 710, Johannesburg
  - Teva Investigational Site 711, Paarl
  - Teva Investigational Site 706, Pretoria
- Spain (4):
  - Teva Investigational Site 336, Alcoy
  - Teva Investigational Site 434, Coslada (Madrid)
  - Teva Investigational Site 433, Vitoria-Gasteiz
  - Teva Investigational Site 430, Vitoria-Gasteiz
- Ukraine (12):
  - Teva Investigational Site 181, Dnipropetrovsk
  - Teva Investigational Site 872, Donetsk
  - Teva Investigational Site 282, Kharkiv
  - Teva Investigational Site 281, Kiev
  - Teva Investigational Site 180, Luhansk
  - Teva Investigational Site 873, Lviv
  - Teva Investigational Site 280, Odesa
  - Teva Investigational Site 875, Odesa
  - Teva Investigational Site 183, Poltava
  - Teva Investigational Site 871, S. Oleksandrivka
  - Teva Investigational Site 184, Simferopol
  - Teva Investigational Site 182, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The final visit of the double-blind study (C10953/3071, /3072, or /3073; NCT01072929, 01072630, or 01305408) serves as the enrollment visit for this study.
Period: Overall Study
Arm/Group | Armodafinil 150-200 mg/Day
Started | 867
Safety Population | 863 (Participants treated)
Full Analysis Population | 859 (Treated participants who had at least 1 post-baseline efficacy assessment.)
Completed | 506 (One participant 'completed' early due to study closeout.)
Not Completed | 361
Not completed — Adverse Event | 63
Not completed — Lack of Efficacy | 35
Not completed — Withdrawal by Subject | 65
Not completed — Protocol Violation | 20
Not completed — Noncompliance with study medication | 12
Not completed — Noncompliance with study procedures | 9
Not completed — Lost to Follow-up | 39
Not completed — Other | 118

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 867
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 525
  Male | 342
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91
  Not Hispanic or Latino | 752
  Unknown or Not Reported | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 118
  White | 709
  More than one race | 0
  Unknown or Not Reported | 28
Weight [Mean (Standard Deviation); unit: kg] | 83.7 (19.75)
Height [Mean (Standard Deviation); unit: cm] | 168.8 (9.54)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (6.43)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: AEs were graded by the investigator for severity on a three-point scale: mild, moderate and severe. Causality is graded as either related or not related. A serious adverse event (SAE) is an AE resulting in death, a life-threatening adverse event, hospitalization, a persistent or significant disability/incapacity, a congenital anomaly/birth defect, or an important medical event that may require medical intervention to prevent any of the previous results.
  Protocol-defined adverse events requiring expedited reporting included skin rash, hypersensitivity reaction, emergent suicidal ideation or suicide attempt, and psychosis.
Time Frame: Day 1 up to Month 6
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 863
participants
  >=1 adverse event | 423
  Severe adverse event | 26
  Treatment-related adverse event | 219
  Deaths | 0
  Other serious adverse events | 27
  Withdrawn from study due to adverse events | 57
  Protocol-defined adverse events | 19

2. Primary Outcome: Participants With Clinically Significant Abnormal Serum Chemistry Values
Description: Summary of serum chemistry tests in which at least one participant had a during study value that was clinically significant abnormal. The test name and criterion for clinically significant abnormal appear in each row.
  * ULN=upper limit of normal
  * BUN=Blood Urea Nitrogen; Uric acid has a normal range of 125-494 μmol/L. Criterion for clinically significant abnormal are different for men and women.
  * GGT = gamma-glutamyl transpeptidase with a normal range of 4-61 U/L
  * ALT = alanine aminotransferase with a normal range of 6-43 U/L
  * BUN = blood urea nitrogen with a normal range of 1.4-8.6 mmol/L
  * AST = aspartate aminotransferase with a normal range of 9-36 U/L
Time Frame: Day 1 to Month 6
Population: Safety population with post-baseline serum chemistry assessments
Measure: Number; unit: participants
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 763
participants
  >=1 clinical significant value | 41
  Uric Acid, M>=625, F>=506 μmol/L | 17
  GGT, >=3*ULN | 16
  ALT, >=3*ULN | 7
  BUN, >=10.71 mmol/L | 7
  AST, >=3*ULN | 3

3. Primary Outcome: Participants With Clinically Significant Abnormal Hematology Values
Description: Summary of hematology tests in which at least one participant had a during study value that was clinically significant abnormal. The test name and criterion for clinically significant abnormal appear in each row.
  * ULN=upper limit of normal
  * WBC - white blood cell counts with a normal range of 3.8-10.7 10^9/L.
  * Hemoglobin with a normal range of 115-181 g/L
  * Hematocrit with a normal range of 0.34-0.54 L/L
  * Platelet counts with a normal range of 130-400 10^9/L
  * ANC= absolute neutrophil counts with a normal range of 1.96-7.23 10^9/L
Time Frame: Day 1 to Month 6
Population: Safety population with post-baseline hematology assessments
Measure: Number; unit: participants
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 757
participants
  >=1 clinical significant value | 13
  WBC, <=3*10^9/L | 5
  Hemoglobin, M<=115, F<=95 g/L | 4
  Hematocrit, M<0.37, F<0.32 L/L | 8
  Platelets, <=75*10^9/L | 1
  ANC, <=1*10^9/L | 2

4. Primary Outcome: Participants With Clinically Significant Abnormal Urinalysis Values
Description: Summary of urinalysis tests in which at least one participant had a during study value that was clinically significant abnormal. Criterion for clinically significant abnormal urinalysis tests was >=2 unit increase from baseline.
Time Frame: Day 1 to Month 6
Population: Safety population with post-baseline urinalysis assessments
Measure: Number; unit: participants
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 761
participants
  >=1 clinical significant value | 28
  Urine hemoglobin | 22
  Urine glucose | 2
  Ketones | 2
  Urine total protein | 2

5. Primary Outcome: Participants With Clinically Significant Abnormal Vital Signs Values
Description: Summary of vital signs tests in which at least one participant had a during study value that was clinically significant abnormal. Criterion for clinically significant abnormal vital signs are based on FDA Neuropharmacological Division criteria:
  * Pulse high: >=120 beats per minute (bpm) and increase of >=15 bpm from baseline
  * Pulse low: <=50 bpm and decrease of >=15 bpm from baseline
  * Sitting systolic blood pressure high: >=180 mm Hg and increase of >=20 mm Hg from baseline
  * Sitting systolic blood pressure low: <=90 mm Hg and decrease of >=20 mm Hg from baseline
  * Sitting diastolic blood pressure high: >=105 mm Hg and increase of >=15 mm Hg from baseline
  * Sitting diastolic blood pressure low: <=50 mm Hg and decrease of >=15 mm Hg from baseline
Time Frame: Day 1 to Month 6
Population: Safety population with post-baseline vital signs assessments
Measure: Number; unit: participants
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 860
participants
  >=1 clinical significant value | 19
  Pulse high | 2
  Pulse low | 2
  Sitting systolic blood pressure high | 3
  Sitting systolic blood pressure low | 8
  Sitting diastolic blood pressure high | 5
  Sitting diastolic blood pressure low | 2

6. Primary Outcome: Change From Baseline to Endpoint in Electrocardiogram (ECG) Values
Description: ECG was conducted at baseline which was before the first dose of study drug in the double-blind study, and at the month-6 visit of the open-label study (or early termination).
  RR= inter-beat intervals
Time Frame: Day 0 (baseline), Month 6 or last post-baseline observation
Population: Safety population of treated participants with both baseline and post-baseline ECG assessments
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 759
msec
  PR interval | 0.2 (16.60)
  QRS interval | 0.0 (7.03)
  QT interval | 1.4 (25.66)
  QTc interval Bazett | 2.2 (19.50)
  QTc interval Fredericia | 1.9 (15.36)
  RR interval | -2.2 (137.98)

7. Primary Outcome: Physical Examination Shifts From Baseline to Endpoint
Description: Baseline is the day prior to double-blind treatment. Assessments are summarized as normal or abnormal. The first assessment is the baseline assessment followed by the endpoint assessment. For example 'normal/abnormal' indicates participants who were normal at baseline and abnormal at endpoint.
  HEENT = Head, Eye, Ear, Nose and Throat exam
Time Frame: Day 0 (baseline), Month 6 (or last post-baseline observation)
Population: Safety population of treated participants with baseline and endpoint assessments Participants n=: General appearance 785, HEENT 784, Chest and lungs 785, Heart 785, Abdomen 785, Musculoskeletal 785, Skin 785, Lymph nodes 780, Neurological 784
Measure: Number; unit: participants
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 863
participants
  General appearance; normal/normal | 714
  General appearance; normal/abnormal | 8
  General appearance; abnormal/normal | 23
  General appearance; abnormal/abnormal | 40
  HEENT: normal/normal | 753
  HEENT: normal/abnormal | 3
  HEENT: abnormal/normal | 15
  HEENT: abnormal/abnormal | 13
  Chest+lungs: normal/normal | 780
  Chest+lungs: normal/abnormal | 0
  Chest+lungs: abnormal/normal | 5
  Chest+lungs: abnormal/abnormal | 0
  Heart: normal/normal | 781
  Heart: normal/abnormal | 2
  Heart: abnormal/normal | 1
  Heart: abnormal/abnormal | 1
  Abdomen: normal/normal | 751
  Abdomen: normal/abnormal | 5
  Abdomen: abnormal/normal | 16
  Abdomen: abnormal/abnormal | 13
  Musculoskeletal: normal/normal | 756
  Musculoskeletal: normal/abnormal | 7
  Musculoskeletal: abnormal/normal | 11
  Musculoskeletal: abnormal/abnormal | 11
  Skin: normal/normal | 707
  Skin: normal/abnormal | 9
  Skin: abnormal/normal | 41
  Skin: abnormal/abnormal | 28
  Lymph nodes: normal/normal | 779
  Lymph nodes: normal/abnormal | 0
  Lymph nodes: abnormal/normal | 0
  Lymph nodes: abnormal/abnormal | 1
  Neurological: normal/normal | 777
  Neurological: normal/abnormal | 2
  Neurological: abnormal/normal | 2
  Neurological: abnormal/abnormal | 3

8. Secondary Outcome: Change From Baseline to Week 1 and Months 1, 2, 4, 6 and Endpoint in the Total Score From the 30-Item Inventory of Depressive Symptomatology-Clinician-Rated (IDS-C30)
Description: The IDS-C30 is a standardized 30-item, clinician-rated scale to assess the severity of a participant's depressive symptoms. Every effort was made to have the same rater evaluate a participant across all visits.
  Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression. Negative change from baseline values indicate improvement in the severity of depression.
  Baseline was the score before the first dose of study drug in the double-blind study.
Time Frame: Day 0 (baseline), Week 1, Months 1, 2, 4, 6 and the last post-baseline assessment)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 859
units on a scale
  Week 1 (837) | -23.7 (12.10)
  Month 1 (793) | -25.8 (11.61)
  Month 2 (716) | -27.6 (11.38)
  Month 4 (578) | -29.2 (11.68)
  Month 6 (503) | -29.7 (12.06)
  Endpoint (857) | -27.5 (13.08)

9. Primary Outcome: Change From Baseline to Endpoint in Body Weight
Description: Baseline was the score before the first dose of study drug in the double-blind study.
Time Frame: Day 0 (baseline), Month 6 (or last post-baseline observation)
Population: Safety population of treated participants with both baseline and post-baseline assessments.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 788
kg | -0.8 (5.67)

10. Primary Outcome: Change From Baseline to Endpoint in the Young Mania Rating Scale (YMRS) Total Score
Description: The YMRS is a clinician-rated, 11-item checklist used to measure the severity of manic episodes. Information for assigning scores is gained from the participant's subjective reported symptoms over the previous 48 hours and from clinical observation during the interview. Seven items are ranked 0 through 4 and have descriptors associated with each severity level. Four items (irritability, speech, content, and disruptive-aggressive behavior) are scored 0 through 8 and have descriptors for every second increment. The total scale is 0-60. A score of ≤12 indicates remission of manic symptoms, and higher scores indicate greater severity of mania. Negative change from baseline scores indicate a decrease in severity of mania.
  Baseline was the score before the first dose of study drug in the double-blind study.
Time Frame: Day 0 (baseline), Month 6 or last post-baseline observation
Population: The safety analysis set includes randomized participants who took 1 or more doses of study drug. The number analyzed includes participants with both baseline (double-blind study) and treatment assessments during the open-label study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 858
units on a scale | -0.7 (4.28)

11. Primary Outcome: Participants With Findings During the Open-Label Study on the Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV)
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The number of participants who had findings on any of the C-SSRS-SLV (SLV=since last visit) categories at any of the time frames are indicated.
  - C-SSRS=Columbia Suicide Severity Rating Scale
Time Frame: Day 1, Week 1, Months 1, 2, 4 and 6 or last post-baseline visit
Population: Safety population; only 19 participants were asked the last three questions as the inclusion of these questions depends on physician assessment.
Measure: Number; unit: participants
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 863
participants
  Suicidal behavior - Actual attempt | 1
  Non-suicidal self-injurious behaviour | 1
  Suicidal behavior - Interrupted attempt | 0
  Suicidal behavior - Aborted attempt | 0
  Suicidal behavior - suicidal behavior | 0
  Suicidal behavior - Preparatory acts/behavior | 1
  Suicidal behavior - Completed suicide | 0
  Suicidal ideation - Wish to be dead | 15
  Non-specific active suicidal thoughts | 4
  Any methods (not plan) w/o intent to act | 2
  Some intent to act, w/o specific plan | 1
  Suicidal ideation - Specific plan and intent | 1

12. Secondary Outcome: Change From Baseline to Week 1 and Months 1, 2, 4, 6 and Endpoint in the Total Score From the 16-Item Quick Inventory of Depressive Symptomatology-Clinician-Rated (QIDS-C16)
Description: The QIDS-C16 was derived from specified items in the IDS-C30, clinician-rated scale to assess the severity of a participant's depressive symptoms. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating the most severe depression. Negative change from baseline values indicate improvement in the severity of depression.
  Baseline was the score before the first dose of study drug in the double-blind study.
Time Frame: Day 0 (baseline), Week 1, Months 1, 2, 4, 6 and the last post-baseline assessment)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 859
units on a scale
  Week 1 (838) | -9.3 (4.68)
  Month 1 (793) | -10.0 (4.47)
  Month 2 (716) | -10.6 (4.52)
  Month 4 (578) | -11.1 (4.70)
  Month 6 (503) | -11.3 (4.69)
  Endpoint (857) | -10.6 (5.07)

13. Secondary Outcome: Change From Baseline to Week 1 and Months 1, 2, 4, 6 and Endpoint in the Clinical Global Impression of Severity (CGI-S) for Depression
Description: The CGI-S is an observer-rated scale that measures illness severity on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). Negative change from baseline values indicate improvement in the severity of depression.
  Baseline was the score before the first dose of study drug in the double-blind study.
Time Frame: Day 0 (baseline), Week 1, Months 1, 2, 4, 6 and the last post-baseline assessment)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 859
units on a scale
  Week 1 (838) | -1.7 (1.17)
  Month 1 (791) | -1.9 (1.17)
  Month 2 (716) | -2.0 (1.18)
  Month 4 (578) | -2.2 (1.16)
  Month 6 (502) | -2.3 (1.18)
  Endpoint (859) | -2.0 (1.31)

14. Secondary Outcome: Change From Baseline to Endpoint in the Global Assessment for Functioning (GAF) Scale
Description: The Global Assessment of Functioning (GAF) is a numeric scale (1 through 100) used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of adults, e.g., how well or adaptively one is meeting various problems-in-living. Ratings of 1 - 10 mean the participant is in persistent danger of severely hurting self or others (e.g., recurrent violence) or persistent inability to maintain minimal personal hygiene or serious suicidal act with clear expectation of death. Ratings of 91 - 100 indicate no symptoms, and the participant exhibits superior functioning in a wide range of activities, life's problems never seem to get out of hand, is sought out by others because of his or her many positive qualities. Positive change from baseline values indicate improvement in functioning.
  Baseline was the score before the first dose of study drug in the double-blind study.
Time Frame: Day 0 (baseline), Month 6 or the last post-baseline assessment)
Population: Full analysis set of participants with both a baseline and post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 779
units on a scale | 17.7 (13.61)

15. Primary Outcome: Change From Baseline to Endpoint in the Insomnia Severity Index (ISI) Total Score
Description: The ISI is a participant-rated, 7-item questionnaire designed to assess the severity of the participant's insomnia. Each item is ranked 0 (none) through 4 (very severe) and has a descriptor associated with each severity level. Total range is 0 (no insomnia) to 28 (very severe insomnia). Responses to each item are added to obtain a total score to determine the severity of insomnia. Negative change from baseline scores indicate a decrease in severity of insomnia. Baseline was the assessment before the first dose of study drug in the double-blind study.
Time Frame: Day 0 (baseline), Month 6 (or last post-baseline observation)
Population: Safety population of treated participants with both a baseline and post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 855
units on a scale | -9.1 (7.66)

16. Primary Outcome: Change From Baseline to Endpoint in the Hamilton Anxiety Scale (HAM-A) Total Score
Description: HAM-A measures the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Negative change from baseline scores indicate a decrease in severity of anxiety.
  Baseline was the score before the first dose of study drug in the double-blind study.
Time Frame: Day 0 (baseline), Month 6 or last post-baseline observation
Population: Safety population of participants with both a baseline and post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil 150-200 mg/Day
Number analyzed (Participants) | 786
units on a scale | -6.2 (5.68)

ADVERSE EVENTS:
Time Frame: Day 1 up to 6 months
Arm/Group | Armodafinil 150-200 mg/Day
Serious Adverse Events (participants affected / at risk) | 27/863
Other Adverse Events (participants affected / at risk) | 133/863
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil 150-200 mg/Day (N=863)
Angina pectoris (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Torsade de pointes (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 3 (3)
Homicidal ideation (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 5 (6)
Suicidal ideation (Psychiatric disorders) | 3 (3)
Suicide attempt (Psychiatric disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil 150-200 mg/Day (N=863)
Headache (Nervous system disorders) | 96 (119)
Insomnia (Psychiatric disorders) | 49 (56)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.